CLINICAL TRIAL: NCT01876992
Title: Pilot Study of Metformin-induced CBP Phosphorylation at the Cellular Level and Corresponding Clinical Dose Response in Adults and Children
Brief Title: Metformin at the Cellular Level and Dosing for Diabetes Mellitus (DM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All investigators/co-investigators relocating to other institutions.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00046072; NA_00046072 (Other: JohnHopkinsU)
Record Dates: First submitted 2013-05-02; First posted 2013-06-13 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Diabetes; Pre-diabetes; Obesity
Keywords: diabetes; pediatrics; obesity; healthy volunteers; metformin; nutrition; healthy controls; bmi
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Obesity | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Doses will be increased incrementally. Decisions to escalate the metformin dose will be made based upon tolerability of side effects as described in the schedule of evaluations to follow. All subjects will be monitored for safety while receiving metformin. Any participant with blood glucose of <60mg/dl at any time while receiving metformin will have therapy stopped and will be withdrawn from the study.
  For children <50kg:
  Baseline:250mg po qd, Week 2:250mg po bid, Week 4:500mg po am/250mg po pm, Week 8:500mg po bid.
  For children ≥50kg:
  Baseline:500mg po qd, Week 2:500mg po bid, Week 4:1000mg po am/500mg po pm, Week 8:1000mg po bid.
  For adults:
  Baseline:500mg po qd,Week2:500mg po bid,Week 4:1000mg po am/500mg po pm,Week 8:1000mg po bid.
  Interventions: Drug: Metformin
- Obese Controls (No Intervention): Three obese but otherwise healthy adult participants will be recruited into the study as controls. These will be individuals who are not currently (or previously) on any diabetic medication including metformin.
  There will be a single study visit and no medication will be administered. They will be administered a meal and pre and post-prandial blood samples will be drawn.

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage, Fortamet
  Arms: Metformin

SUMMARY:
The investigators know that metformin works at the level of the cells in the body by acting on a protein called Cyclic amine monophosphate- Response Binding Elements (CREB) binding protein or Constitutive Reverter of eIF2α Phosphorylation (CREP) Binding Protein (CBP). What the investigators do not know is how this process is affected when the dose of the metformin is increased or changed.

Currently the same doses of metformin are often used in both children and adults, but it is possible that the dose of metformin should be based on age and weight. Understanding how CBP works could potentially help us to tailor metformin treatment individually for patients based on their age, weight and CBP response.

DETAILED DESCRIPTION:
Our studies have shown that metformin acts at the cellular level by acting on a target protein, Cyclic amine monophosphate-Response Binding Elements (CREB) binding protein or CREP Binding Protein (CBP). Patients are treated with many different doses of metformin, some patients respond well to low doses while others require much higher doses. The investigators do not understand why this may be and are interested in knowing if the investigators can treat patents effectively with low doses. What the investigators do not know is how this process is affected when the dose of the metformin is increased or changed. Changes in metformin's target protein will provide evidence on the effectiveness of the dose.

Also, currently the same doses of metformin are often used in both children and adults, but it is possible that the dose of metformin should be based on age and weight. Understanding how CBP works could potentially help us to tailor metformin treatment individually for patients based on their age, weight and CBP response.

ELIGIBILITY:
Pediatric Inclusion Criteria:

* Children 10-17 years.
* Both genders (male and female)
* All children must have a Primary Care Physician and/or an Endocrinologist who must be aware that the child under their care will be part of the study.
* All children must have a Primary Care Physician and/or an Endocrinologist who is considering initiating metformin therapy now or in the near future as part of standard clinical care.
* Naïve to metformin.
* Either: Prediabetic children Or diabetic children under good glycemic control

Pediatric Exclusion Criteria:

* Children ages 10-17 who do not have parental consent and/or do not give assent
* Children living in foster care
* Children with allergies to foods in the breakfast menu
* Children who currently consume any alcohol
* Children on current antidiabetic medication or those who have been on any antidiabetic medication in the 3 months prior to enrolment
* Children with a history of /or concurrent chronic disease (eg. heart, kidney, liver disease or any type of malignancy or pre-malignant condition) that required hospitalization within the last 6 months
* Pregnancy
* Refusal by a female participant who is of child bearing potential and sexually active to use contraceptive methods such as oral contraceptive pills, barrier methods and abstinence
* Children weighing less than 36 kg
* Children with any condition that increases the risk of lactic acidosis (e.g. cancer, infection, congestive heart failure, renal disease )
* Children with history of recent hospitalization for surgery, dehydration, sepsis, hypoxemia (within the past 6 months)
* Children with history of weight loss, polyuria and polydipsia
* Children who are currently enrolled in a weight management program
* Children with known hypersensitivity to metformin
* Children with a fasting blood glucose of >180mg/dl
* Children with a HbA1c level of ≥7%
* Children with glycosuria
* Children with clinical or laboratory evidence of hepatic disease- transaminase levels three times the upper normal range (Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT)) and/or a increased level of Gamma-glutamyltransferase (GGT), Prothrombin Time (PT), International Normalized Ratio (INR) from the reference normal range and a serum albumin less than the reference normal range of the Johns Hopkins Clinical Laboratories.
* If iodinated contrast is used on a participant, due to possible acute alteration of renal function resulting in increased risk of lactic acidosis, the participant will be excluded.
* Children with renal impairment

  * In children >50kg, renal impairment is defined by a serum creatinine 1.4 mg/dl or higher in females or 1.5mg/dl or higher in males OR estimated Glomerular Filtration Rates (eGFR) ≤60mL/min by the Schwartz formula.
  * In children <50kg, renal impairment is defined by eGFR <100 mL/min by the Schwartz formula.
* Children with acid-base disturbance as defined by serum bicarbonate levels less than 20mEq/L or greater than 29mEq/L.

Adult Inclusion Criteria:

* Adults 18-79 years
* Both genders (male and female)
* All participants must have a Primary Care Physician and/or an Endocrinologist who must be aware that the adult under their care will be part of the study
* All participants must have a Primary Care Physician and/or an Endocrinologist who is considering initiating metformin therapy now or in the near future as part of standard clinical care.
* Naive to metformin
* EITHER: Prediabetic adults OR diabetic adults, under fair glycemic control:

Adult Exclusion Criteria:

* Pregnancy
* Adults who are not able to understand the Informed Consent document and who are unwilling to do the study
* Adults with allergies to any of the foods in the breakfast menu
* Adults on current antidiabetic medication or on any antidiabetic medication in the 3 months prior to enrolment.
* Adults with a history of /or concurrent chronic disease (e.g. heart, kidney, liver disease or any type of malignancy or pre-malignant condition) that required hospitalization within the last 6 months
* Refusal by a female participant who is of child bearing potential and sexually active to use contraceptive methods such as oral contraceptive pills, barrier methods and abstinence
* Adults with excessive current intake of alcohol (>2 drinks/day for males and >1 drink/day for females)
* Adults who have engaged in binge drinking (>5 drinks within a 2 hour period) in the last 3 months
* Adults with history of recent hospitalization for surgery, dehydration, sepsis, hypoxemia (past 6 months)
* Hypersensitivity to metformin.
* Adults with fasting blood glucose of >180mg/dl.
* Adults with HbA1c level of ≥8%
* Adults with glycosuria.
* Adults with any condition that increases the risk of lactic acidosis (e.g. cancer, infection, congestive heart failure, renal disease )
* Adults with clinical or laboratory evidence of hepatic disease- transaminase levels three times the upper normal range (AST and ALT) and/or a increased level of GGT, PT, INR from the reference normal range and a serum albumin less than the reference normal range of the Johns Hopkins Clinical Laboratories.
* If iodinated contrast is used on a participant, due to possible acute alteration of renal function resulting in increased risk of lactic acidosis, the adult participant will be excluded.
* Adults with renal impairment as defined by a serum creatinine 1.4 mg/dl or higher in females or 1.5mg/dl or higher in males OR estimated Glomerular Filtration Rates (eGFR) ≤60mL/min by Modification of Diet in Renal Disease (MDRD) formula.
* Adults with acid-base disturbance as defined as serum bicarbonate levels less than 20mEq/L or greater than 29mEq/L.

Adult Obese Control Inclusion Criteria:

* Age 18-79
* Both genders (male and female)
* BMI > 30 kg/m2

Adult Obese Control Exclusion Criteria:

* Subjects previously or currently on any diabetes medication, including metformin, will be excluded.
* Pregnancy
* Subjects with history of or concurrent chronic disease (e.g. heart, kidney, liver disease or any type of malignancy or pre-malignant condition) that required hospitalization within the last 6 months will be excluded.
* Adults with allergies to any of the foods in the breakfast menu
* Adults with excessive current intake of alcohol (>2 drinks/day for males and >1 drink/day for females)
* Adults who have engaged in binge drinking (>5 drinks within a 2 hour period) in the last 3 months

Ages: 10 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally Radovick, MD, Principal Investigator — Johns Hopkins University Department of Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited through the Clinical Research Center.
Groups:
- Metformin: Doses will be increased incrementally. Decisions to escalate the metformin dose will be made based upon tolerability of side effects as described in the schedule of evaluations to follow. All subjects will be monitored for safety while receiving metformin. Any participant with blood glucose of <60mg/dl at any time while receiving metformin will have therapy stopped and will be withdrawn from the study.
  For children <50kg:
  Baseline:250mg po qd, Week 2:250mg po bid, Week 4:500mg po am/250mg po pm, Week 8:500mg po bid.
  For children ≥50kg:
  Baseline:500mg po qd, Week 2:500mg po bid, Week 4:1000mg po am/500mg po pm, Week 8:1000mg po bid.
  For adults:
  Baseline:500mg po qd,Week2:500mg po bid,Week 4:1000mg po am/500mg po pm,Week 8:1000mg po bid.
  Metformin
Period: Overall Study
Arm/Group | Metformin | Obese Controls
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metformin: Doses will be increased incrementally. Decisions to escalate the metformin dose will be made based upon tolerability of side effects as described in the schedule of evaluations to follow. All subjects will be monitored for safety while receiving metformin. Any participant with blood glucose of <60mg/dl at any time while receiving metformin will have therapy stopped and will be withdrawn from the study.
  For children <50kg:
  Baseline:250mg po qd, Week 2:250mg po bid, Week 4:500mg po am/250mg po pm
  , Week 8:500mg po bid.
  For children ≥50kg:
  Baseline:500mg po qd, Week 2:500mg po bid, Week 4:1000mg po am/500mg po pm, Week 8:1000mg po bid.
  For adults:
  Baseline:500mg po qd,Week2:500mg po bid,Week 4:1000mg po am/500mg po pm,Week 8:1000mg po bid.
  Metformin
- Total: Total of all reporting groups
Arm/Group | Metformin | Obese Controls | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 32 [19 to 44] | 36 [22 to 38] | 34 [19 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: % Cyclic Amine Mono Phosphate (cAMP) Response Element Binding Protein (CBP) White Blood Cell (WBC) Phosphorylation (Metformin Treated vs no Treatment)
Description: To assess metformin-induced Cyclic Amine Mono Phosphate (cAMP) response element binding protein (CBP) phosphorylation in circulating white blood cells both in vivo and ex vivo and determine its relationship to subsequent changes in body mass index, fasting blood glucose.
Time Frame: 10 weeks
Measure: Mean (Full Range); unit: percent phosphorylation
Arm/Group | Metformin | Obese Controls
Number analyzed (Participants) | 5 | 5
percent phosphorylation | 15 [11 to 18] | 9 [6 to 12]

2. Secondary Outcome: Change in BMI
Description: The BMI is an index measure of body weight and is used to define states of obesity. Height ( in meters) and weight (in Kilograms) are used to calculate a BMI (kg/m2).
Time Frame: Baseline and after about 30 days
Measure: Mean (Full Range); unit: change in BMI (kg/m2)
Arm/Group | Metformin | Obese Controls
Number analyzed (Participants) | 5 | 5
change in BMI (kg/m2) | -0.5 [-0.9 to 0.2] | 0 [-0.3 to 0.2]

3. Secondary Outcome: Fasting Blood Glucose.
Description: A fasting blood sugar level less than 100 mg/dL is normal. A fasting blood sugar level from 100 to 125 mg/dL is considered prediabetes. If a subject has a blood sugar of 126 mg/dL or higher on two separate tests, they are diagnosed with diabetes. Metformin decreases fasting blood sugar.
Time Frame: 30 days
Population: Data were not collected for this outcome measure.
Arm/Group | Metformin | Obese Controls
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Effect of Dose Escalation
Description: Compare the effect of dose escalation of metformin on CBP phosphorylation in white blood cells in both in vivo and ex vivo assays to subsequent physiological changes in vivo for adults and children. CBP phosphorylation will be measured by western blot analysis using a probe that is specific for the phosphorylated CBP protein. The outcome will be the % difference between the patient before starting metformin and at each dose increment.
Time Frame: Approximately Week 10
Population: Escalating CBP phosphorylation was measured.
Measure: Mean (Full Range); unit: percent phosphorylation
Arm/Group | Metformin | Obese Controls
Number analyzed (Participants) | 5 | 5
percent phosphorylation | 21 [15 to 25] | 8 [6 to 10]

ADVERSE EVENTS:
Arm/Group | Metformin | Obese Controls
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes